CLINICAL TRIAL: NCT05984979
Title: The Daytime Circadian Rhythm in Exhaled Volatile Organic Compounds in People Living Without and With Type 1 and 2 Diabetes: an Exploratory Study
Brief Title: The Daytime Circadian Rhythm in Exhaled Volatile Organic Compounds in People Living Without and Diabetes
Acronym: VOCircle
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); DCB Research AG (Other)
Responsible Party: Sponsor
Other Study IDs: VOCircle
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — The spare aliquots used for the study research will be destroyed after the completion of the study. Purified oral and gut microbiota DNA will be stored up to 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People without diabetes
  Interventions: Other: Standardized meal
- People with type 1 diabetes
  Interventions: Other: Standardized meal
- People with type 2 diabetes
  Interventions: Other: Standardized meal

INTERVENTIONS:
Other: Standardized meal — The participants will receive a standardized meal for breakfast

SUMMARY:
Exhaled volatile organic compounds will be measured during daytime with the goal to identifying circadian variability. The study incudes three subgroups: people without diabetes, people with type 1 diabetes, and people with type 2 diabetes. A total of 60 people will be recruited for the study.

ELIGIBILITY:
Inclusion criteria

Subgroup 1:

* Age 18 or older
* HbA1c below 6.5%
* Written informed consent

Subgroup 2:

* Age 18 or older
* T1D (Type 1 diabetes) with MDI (multiple daily injection) or CSII (Continuous subcutaneous insulin infusion therapy) therapy >1 year
* Written informed consent

Subgroup 3

* Age 18 or older
* T2D (Type 2 diabetes) with oral antidiabetic medication or insulin therapy
* Written informed consent

Exclusion criteria

* Pregnancy or breastfeeding
* Smoking (last cigarette less than 6 months ago)
* Any chronical lung and intestinal disease diagnosis (such as intestinal bowel disease (IBD); asthma; COPD (chronic obstructive pulmonary disease); lung cancer, …)
* Coeliac disease
* Lactose and fructose intolerance
* Any acute disease diagnosis (such as viral or bacterial infection)
* Drinking habit of more than four units of alcohol per day
* Current inhaled medicines treatments
* Antibiotic treatment in the previous 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 participants with the following subgroups: Subgroup 1: People without diabetes Subgroup 2: People diagnosed with T1D Subgroup 3: People diagnosed with T2D
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
VOC Patterns over time as gallery plots | During the study procedure (approximately 8 hours)
  Gallery plots (3D visualization of retention index, drift time, ion current) from selected VOC peaks over time.
VOC Patterns over time as boxplots | During the study procedure (approximately 8 hours)
  Box plots from selected VOC peaks over time.

SECONDARY OUTCOMES:
Capillary blood glucose | During the study procedure (approximately 8 hours)
  Correlation between capillary blood glucose and VOCs
Correlation between VOCs in breath intestinal microbiota | day 1
  Correlation between VOCs in breath and intestinal microbiota species abundance
Correlation between VOCs in breath oral microbiota | day 1
  Correlation between VOCs in breath and oral microbiota species abundance
Correlation between VOCs and subgroups | day 1 or 8 hours
  Wilcoxon signed-rank test will be used to explore if the patterns in VOCs differ between subgroup: people without diabetes, people living with T1D, and people living with T2D

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Witthauer, Prof.Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No